CLINICAL TRIAL: NCT02328417
Title: Enhanced Recovery After Radical Cystectomy Study
Status: Completed | Type: Observational
Sponsor: Carlos Llorente (Other)
Responsible Party: Sponsor-Investigator, Carlos Llorente, Doctor in Medicine, Hospital Universitario Fundación Alcorcón
Organization: Hospital Universitario Fundación Alcorcón (Other)
Other Study IDs: PRO-RAC
Record Dates: First submitted 2014-11-18; First posted 2014-12-31 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Consecutive radical cystectomies up to 94 patients in 13 participating hospitals in Madrid, Spain. These patients will be taken care of as it is done regularly in each of participating hospitals. All study variables will be prospectively collected in this group
- Active Treatment: After recruiting cotrol group, another consecutive radical cystectomies up to 94 patients in 13 participating hospitals will be recruited and the following measures will be followed with them:
  I.-PREOPERATIVE MEASURES: (eight measures according to Protocol) II.- INTRAOPERATIVE MEASURES: (six measures according to Protocol) III.- POSTOPERATIVE MEASURES: (eight measures according to Protocol)
  Interventions: Other: Consecutive radical cystectomies

INTERVENTIONS:
Other: Consecutive radical cystectomies — Pre-, intra- and post-operative clinical measures during radical cystectomy clinical process
  Groups: Active Treatment

SUMMARY:
Prospective non randomized study of two cohorts: usual protocol and the application of accelerated recovery protocol. F/up after discharge, 90 days and thereafter according to protocol of each center. Compliance to be assessed.

DETAILED DESCRIPTION:
This is a prospective non randomized study of two cohorts, one defined by the usual protocol and the other one by the application of accelerated recovery protocol. It's discarded a priori a prospective randomized trial, since it does not seem feasible to avoid byass of control group when synchronizing the active intervention and control. Subjects surgery will be followed after discharge for a minimum of 90 days, and thereafter according to protocol of each center. Patients will be provided with a satisfaction survey 90 days after surgery.

The degree of compliance with the protocol will be assessed through a checklist indicating compliance with each of the steps of the protocol in both groups. All patients will sign an informed consent for the study authorizing the use of their clinical data for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for radical cystectomy in the participating hospitals
* Signed informed consent

Exclusion Criteria:

* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive male and female patients older than 18 years submitted to radical cystectomy due to bladder cancer in the 13 participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
In-hospital length-of-stay (LOS), defined as the number of days since the admission of the patient to the hospital until the day of discharge, Morbidity of surgery. Categorized by the Clavien complications scale at 30-, 60- and 90-postoperative days | 5-40 days
  Day 1: Admission to the hospital Last day of accountant: Discharge from the hospital or death in the hospital.

SECONDARY OUTCOMES:
Mortality at 30-, 60- and 90- postoperative days | 90 days
30-day readmission rate | 30 days
Transfusion rate | 90 days
Patient satisfaction measured with the enclosed questionnaire | 90 days
  Do you know the names of your attending physician and nurse?
  The quality of the preoperative care and information has been:
  The quality of the postoperative care and information has been:
  Do you think that the information on the care of your urostomy has been enough? Yes/No If NO, on which of the following points would you have liked receiving more information? Types of collecting bags and accessories Stomal hygiene and change of bags Complications of the stoma and the surrounding skin Counseling on food habits, dress apparel, and physical and sexual activity Comunity counselling: Stoma therapist, patients associations If you had a neobladder performed, were you trained in self-catheterization ? How would you rate your motivation in learning the above mentioned issues?
  In all, the quality of the health care that you have received is:

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Llorente, MD, Principal Investigator — Hospital Fundación de Alcorcón
Locations (12):
- Spain (12):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid